CLINICAL TRIAL: NCT01921062
Title: Kinesthetic Motor Imagery Training During Immobilization to Improve Wrist Functional Outcome After a Distal Radius Fracture in Women of 45-75 Years of Age
Brief Title: Motor Imagery in Rehabilitation After a Distal Radius Fracture
Acronym: MIDRF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Severe difficulties with recruiting participants
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, D.C. Broekstra, MSc, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIDRF; NL36638.042.11 (Other: Central Committee on Research Involving Human Subjects)
Record Dates: First submitted 2013-08-07; First posted 2013-08-13 (Estimated); Results first posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-07

CONDITIONS: Distal Radius Fracture
Keywords: Distal radius fracture; Motor imagery; Immobilisation; Effectivity
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients allocated to the control group only receive standard treatment.
- Motor imagery (Experimental): Patients allocated to this arm perform kinesthetic motor imagery during the immobilisation period.
  Interventions: Behavioral: Motor imagery

INTERVENTIONS:
Behavioral: Motor imagery — The kinesthetic motor imagery training consists of the imagination of flexion, extension, abduction, adduction, pronation and supination of their injured wrist.
  Arms: Motor imagery

SUMMARY:
The aim of this study is to determine whether motor imagery training during the immobilisation period in patients with a distal radius fracture, results in an improved functional outcome compared to patients who do not perform motor imagery.

DETAILED DESCRIPTION:
Rationale: Distal radius fracture (DRF) is a common injury that may lead to prolonged function restrictions, decreased range of motion, reduced grip strength and pain. These symptoms may be caused by physical changes due to the injury and/or by the 4-6 weeks immobilization that is part of the conservative treatment. However, it might also be that neural changes during the immobilization play an important role. Such changes might be prevented by motor imagery training during the immobilization period. So, when neural changes are prevented, this may lead to a better functional outcome.

Objective: The objective is to improve the functional outcome in distal radius fracture patients, specified as an increase in function, dexterity, grip strength, range of motion, and decrease of pain.

Study design: Parallel group randomized controlled trial, with a post-test only control group design. Patients in the experimental group perform motor imagery training during the immobilization period, in addition to the regular treatment. Patients in the control group receive regular treatment.

Study population: Female DRF-patients who are conservatively treated by a cast, aged 45-75 years. The fracture must be a low energy trauma caused by a fall. Patients with a score higher than 72 on the Vividness of Motor Imagery Questionnaire (VMIQ) are excluded, as well as patients with co-morbidities that might influence the wrist function, or motor imagery-ability, and patients with no understanding of Dutch language. The patients are randomly allocated to the experimental or control group by restricted randomization to ensure equal group sizes.

Intervention: Motor imagery training during the immobilization period).

Main study parameters/endpoints: The main study parameter is function. Secondary study parameters are dexterity, range of motion, grip strength, and pain.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* non-comminutive distal radius fracture
* 45 to 75 years of age

Exclusion Criteria:

* distal radius fracture caused by HET
* comorbidities possibly influencing wrist function
* comorbidities possibly influencing motor imagery ability
* score higher than 72 on the Vividness of Motor Imagery Questionnaire

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin W. Stenekes, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
No plan currently available, but we are open for collaborations.

REFERENCES:
- [Result] Broekstra DC, Mouton LJ, van der Sluis CK, IJpma FFA, Stenekes MW. Hand function in patients with distal radius factures after home-based kinaesthetic motor imagery training. J Hand Surg Eur Vol. 2022 Jun;47(6):656-658. doi: 10.1177/17531934221075945. Epub 2022 Feb 1. No abstract available. PMID 35102780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited through invitation letter after ER visit. Recruitment took place between July 2011 and January 2020
Pre-assignment Details: Out of 117 patients, 3 did not respond to the invitation and 42 responded that they did not want to participate
Period: Overall Study
Arm/Group | Control | Motor Imagery
Started | 28 | 38
Completed | 19 | 22
Not Completed | 9 | 16
Not completed — Withdrawal by Subject | 0 | 7
Not completed — Adverse Event | 5 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — VMIQ score > 72 | 4 | 1
Not completed — Logistic error | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Motor Imagery | Total
Number analyzed (Participants) | 19 | 24 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (6.7) | 58.7 (7.5) | 58.7 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 19 | 24 | 43
Fracture type (extra-articular) [Count of Participants; unit: Participants] | 16 | 18 | 34
AO classification [Count of Participants; unit: Participants] — Fracture type in terms of AO classification for the distal radius (code 23), being classified as extra-articular (A), partial articular (B), or intra-articular (C)
  Participants
    23A | 14 | 16 | 30
    23B | 2 | 2 | 4
    23C | 3 | 6 | 9
Dominant hand affected [Count of Participants; unit: Participants] | 10 | 18 | 28
Hand dominance [Count of Participants; unit: Participants]
  Right | 17 | 21 | 38
  Left | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Hand Function
Description: Self-perceived hand function (construct) measured using the Patient Rated Wrist Hand Evaluation (PRWHE, scale). The score can range between 0 (no functional complaints) to 100 (unable to function)
Time Frame: 2 days after cast removal
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Motor Imagery
Number analyzed (Participants) | 15 | 20
score on a scale | 44.3 (19.4) | 48.0 (23.2)

2. Other Pre Specified Outcome: Grip Strength (Difference Unaffected - Affected)
Description: Four different strength measurements were assessed; power grip, three-jaw chuck pinch, key pinch, and two-point pinch (Mathiowetz et al., 1984), using a digital Jamar dynamometer and pinch grip meter (H500 Hand Kit, Biometrics Ltd., Newport, United Kingdom), expressed in kilograms. Grip and pinch strength of the non-affected hand were measured as reference. The averages of three measurements were used in all analyses.
Time Frame: 2 weeks after cast removal
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Control | Motor Imagery
Number analyzed (Participants) | 19 | 22
kg
  Power grip | 11.5 (5.0) | 10.5 (5.8)
  Key pinch | 2.2 (1.5) | 1.7 (1.2)
  Three-jaw pinch | 2.4 (1.5) | 2.2 (1.4)
  Two-point pinch | 1.4 (1.1) | 1.0 (1.2)

3. Other Pre Specified Outcome: Dexterity
Description: Dexterity (construct) as measured using the Sequential Occupational Dexterity Assessment (SODA, scale). The SODA is a valid and reliable instrument that measures bimanual dexterity during activities of daily living (van Lankveld et al. 1996). The SODA consists of 12 tasks, and it takes 20 minutes to complete it. The performance on the tasks is scored by the experimenter. The score for each task is build up by two different components. One component concerns how the task is performed, and the other component concerns the difficulty the patient experiences during the execution of the task. For some tasks, only one hand is scored, while for other tasks both hands are scored. The final score ranges from 0-108, where 0 means that the patient is unable to perform any of the tasks, and 108 means that all tasks were performed as requested without any difficulty (van Lankveld et al. 1996).
Time Frame: Directly after cast removal
Population: Not all patients were able to perform the tasks of the SODA, explaining lower number of participants included in the analysis
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Motor Imagery
Number analyzed (Participants) | 17 | 16
score on a scale | 87.5 [72.3 to 92] | 88.0 [77.0 to 95.0]

4. Other Pre Specified Outcome: Current Pain Level
Description: Current pain level, measured using a Visual Analogue Scale (VAS), 0 (best) - 100 (worst)
Time Frame: Directly after cast removal
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Motor Imagery
Number analyzed (Participants) | 19 | 23
score on a scale | 10.0 [2.5 to 23.5] | 4.0 [2.0 to 18.0]

5. Other Pre Specified Outcome: Pain Relief
Description: Current pain relief, measured using a Visual Analogue Scale (VAS), 0 (worst) - 100 (best)
Time Frame: Directly after cast removal
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Motor Imagery
Number analyzed (Participants) | 19 | 23
score on a scale | 69.0 [48.0 to 90.5] | 78.0 [49.0 to 90.0]

6. Other Pre Specified Outcome: Range of Motion
Description: Active range of motion (flexion, extension, radial deviation, ulnar deviation, pronation and supination)(Gajdosik and Bohannon, 1987) was measured in degrees once using a digital goniometer (R500 Range of Motion Kit, Biometrics Ltd., Newport, United Kingdom). ROM of the non-affected hand was also measured as reference.
Time Frame: Directly after cast removal.
Population: Some participants could not do all movements, which explains that some ROMs have a lower number of participants in the analysis
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control | Motor Imagery
Number analyzed (Participants) | 21 | 19
degrees
  Extension | 34.7 (13.8) | 25.7 (17.3)
  Flexion | 39.0 (12.2) | 35.8 (20.6)
  Pronation: number analyzed (Participants) | 21 | 18
  Pronation | 8.3 (19.8) | 11.5 (14.0)
  Supination: number analyzed (Participants) | 21 | 18
  Supination | 24.3 (21.5) | 26.4 (25.7)
  Radial deviation | 5.9 (6.6) | 7.1 (7.5)
  Ulnar deviation | 8.5 (6.2) | 13.0 (8.1)

7. Other Pre Specified Outcome: Hand Function
Description: as for outcome 1
Time Frame: 2 weeks after cast removal
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Motor Imagery
Number analyzed (Participants) | 19 | 20
score on a scale | 32.4 (19.2) | 35.3 (20.7)

8. Other Pre Specified Outcome: Grip Strength
Description: as for outcome 2
Time Frame: Directly after cast removal
Population: Not all participants were able to perform the grips or pinch movements requested, explaining why some outcome measures have less patients included in the analysis
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Control | Motor Imagery
Number analyzed (Participants) | 18 | 21
kg
  Power grip: number analyzed (Participants) | 16 | 21
  Power grip | 15.6 (3.6) | 15.2 (5.7)
  Key pinch | 2.9 (1.3) | 2.6 (1.2)
  Three-jaw pinch: number analyzed (Participants) | 17 | 21
  Three-jaw pinch | 3.4 (1.2) | 3.6 (1.7)
  Two-point pinch: number analyzed (Participants) | 17 | 21
  Two-point pinch | 1.9 (0.9) | 2.2 (1.0)

9. Other Pre Specified Outcome: Dexterity
Description: as for outcome 3
Time Frame: 2 weeks after cast removal
Population: Some participants dropped out between T1 and T2
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Control | Motor Imagery
Number analyzed (Participants) | 15 | 18
points | 102.0 [97.5 to 103.5] | 99.5 [92.3 to 105.0]

10. Other Pre Specified Outcome: Current Pain Level
Description: Current pain level, measured using a Visual Analogue Scale (VAS), 0 (best) - 100 (worst)
Time Frame: 2 weeks after cast removal
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Motor Imagery
Number analyzed (Participants) | 19 | 22
score on a scale | 9.0 [3.0 to 13.5] | 8.5 [3.3 to 15.3]

11. Other Pre Specified Outcome: Pain Relief
Description: Current pain relief, measured using a Visual Analogue Scale (VAS), 0 (worst) - 100 (best)
Time Frame: 2 weeks after cast removal
Population: Some participants dropped out between T1 and T2
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control | Motor Imagery
Number analyzed (Participants) | 19 | 22
score on a scale | 67.0 [35.0 to 81.0] | 81.5 [37.0 to 86.3]

12. Other Pre Specified Outcome: Range of Motion
Description: as for outcome 6
Time Frame: 2 weeks after cast removal.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control | Motor Imagery
Number analyzed (Participants) | 19 | 22
degrees
  Extension: number analyzed (Participants) | 18 | 22
  Extension | 18.1 (15.9) | 14.3 (13.0)
  Flexion | 16.2 (21.6) | 21.5 (15.3)
  Pronation: number analyzed (Participants) | 19 | 21
  Pronation | 4.4 (11.9) | 2.5 (13.2)
  Supination: number analyzed (Participants) | 19 | 21
  Supination | 17.5 (21.9) | 20.5 (23.0)
  Radial deviation | 2.7 (5.4) | 4.4 (6.7)
  Ulnar deviation | 9.3 (6.3) | 8.0 (7.9)

ADVERSE EVENTS:
Time Frame: 2 months
Description: Non-fusion of a fracture after 5 weeks of immobilisation
Arm/Group | Control | Motor Imagery
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/24
Other Adverse Events (participants affected / at risk) | 0/19 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=19) | Motor Imagery (N=24)
Non-fusion of conservatively treated distal radius fracture (Musculoskeletal and connective tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The SODA scores appeared to be very much influenced by hand dominance, because of the nature of the activities assessed in the SODA. We therefore decided not to statistically test the SODA scores, but only provide descriptive statistics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT01921062/Prot_SAP_000.pdf